CLINICAL TRIAL: NCT03962803
Title: A Prospective Study on the Immunogenicity and Persistence of Hepatitis B Vaccine in HIV-Infected Patients
Brief Title: Immunogenicity and Persistence of Hepatitis B Vaccination in HIV-Infected Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanxi Medical University (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Suping Wang, Professor, Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018ZX10721202001002001
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Hepatitis B Vaccine
Keywords: Hepatitis B Vaccine; Randomized Controlled Trial; HIV-Infected Patients; Immunogenicity; Long-term Immune Response
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20 µg at months 0, 1, and 6 (Experimental): 20 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6
  Interventions: Biological: 20 µg recombinant hepatitis B vaccine at months 0, 1, and 6
- 20 µg at months 0, 1, 2,and 6 (Experimental): 20 µg recombinant hepatitis B vaccine with four injections at months 0, 1, 2, and 6
  Interventions: Biological: 20 µg recombinant hepatitis B vaccine at months 0, 1, 2, and 6
- 60 µg at months 0, 1, 2,and 6 (Experimental): 60 µg recombinant hepatitis B vaccine with four injections at months 0, 1, 2, and 6
  Interventions: Biological: 60 µg recombinant hepatitis B vaccine at months 0, 1, 2, and 6

INTERVENTIONS:
Biological: 20 µg recombinant hepatitis B vaccine at months 0, 1, and 6 — three-dose, 20 µg per dose
  Arms: 20 µg at months 0, 1, and 6
Biological: 20 µg recombinant hepatitis B vaccine at months 0, 1, 2, and 6 — four-dose, 20 µg per dose
  Arms: 20 µg at months 0, 1, 2,and 6
Biological: 60 µg recombinant hepatitis B vaccine at months 0, 1, 2, and 6 — four-dose, 60 µg per dose
  Arms: 60 µg at months 0, 1, 2,and 6

SUMMARY:
At present, HIV-Infected Patients of Hepatitis B Vaccination in are vaccinated with hepatitis B vaccine according to the standard three-dose schedule immunization program, and the effect of preventing HBV infection is not ideal.

This is a randomized, controlled trial. The study will evaluate the immunogenicity and persistence of 20 µg and 60 µg recombinant hepatitis B vaccine with three or four injections at months 0, 1, and 6 or 0, 1,2, and 6 in HIV-Infected Patients

DETAILED DESCRIPTION:
Participants are randomized in a ratio of 1:1:1 into 20 µg recombinant hepatitis B vaccine group at months 0, 1, and 6 or 20µg recombinant hepatitis B vaccine group at months 0, 1, 2, and 6 or 60µg recombinant hepatitis B vaccine group at months 0, 1, 2, and 6. HBsAg and anti-HBs will be tested during the study period. Adverse reactions will be recorded after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Serologically negative for hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (anti-HBs) and hepatitis B core antibody (anti-HBc) at enrollment
* Sign informed consent, willing to participate in this study

Exclusion Criteria:

* Being pregnant
* Intolerance or allergy to any component of the vaccine
* Any vaccination during the month preceding enrollment
* CD4 cell count ≤ 200 cells/µL
* Patients with severe acute or chronic diseases (such as liver disease, blood disease, cancer), acute onset of chronic diseases and fever
* The use of immunosuppressive agents in patients with nearly three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-06-05 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Anti-HBs Seroconversion Rate at Month 7 | Month 7
  Anti-HBs Seroconversion Rate at month 7 as measured by CMIA

SECONDARY OUTCOMES:
Anti-HBs concentration at month 7 | Month 7
  Anti-HBs concentration at month 7 as measured by CMIA
Occurrence of Adverse Events After Vaccination | Within 7 days after the vaccination
  Occurrence of adverse reactions within 7 days after vaccination with the hepatitis
Anti-HBs Seroconversion Rate at month 12 | Month 12
  Anti-HBs Seroconversion Rate at month 12 as measured by CMIA
Anti-HBs concentration at month 12 | Month 12
  Anti-HBs concentration at month 12 as measured by CMIA
Anti-HBs Seroconversion Rate at month 18 | Month 18
  Anti-HBs Seroconversion Rate at month 18 as measured by CMIA
Anti-HBs concentration at month 18 | Month 18
  Anti-HBs concentration at month 18 as measured by CMIA
Anti-HBs Seroconversion Rate at month 30 | Month 30
  Anti-HBs Seroconversion Rate at month 30 as measured by CMIA
Anti-HBs concentration at month 30 | Month 30
  Anti-HBs concentration at month 30 as measured by CMIA
Anti-HBs Seroconversion Rate at month 42 | Month 42
  Anti-HBs Seroconversion Rate at month 42 as measured by CMIA
Anti-HBs concentration at month 42 | Month 42
  Anti-HBs concentration at month 42 as measured by CMIA

CONTACTS AND LOCATIONS:
Overall Officials: Suping Wang, PhD, Principal Investigator — Shanxi Medical University
Locations (1):
- Shanxi Center for Disease Control and Prevention, Taiyuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng Y, Chen Z, Xie R, Yao T, Wu Y, Yang F, Yuan C, Nie X, Wang F, Liang X, Wang S. Immunogenicity and safety of 4 intramuscular standard-dose and high-dose hepatitis B vaccine in people living with HIV: a randomized, parallel-controlled trial. Expert Rev Vaccines. 2022 Jun;21(6):861-868. doi: 10.1080/14760584.2022.2056024. Epub 2022 Apr 1. PMID 35312441